CLINICAL TRIAL: NCT01326273
Title: Adoptive Transfer of Autologous CMV Specific CD8+ T Cells After Allogeneic Stem Cell Transplantationas Treatment for CMV Reactivation: A Phase I/II Clinical Trial.
Brief Title: Autologous Cytomegalovirus (CMV) Specific CD8+ T Cells as Treatment for CMV Reactivation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JROHH0202
Record Dates: First submitted 2011-03-22; First posted 2011-03-30 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2012-03

CONDITIONS: CMV Reactivation; Allogeneic Stem Cell Transplantation; Autologous CMV Specific CD8+ T Cells
Keywords: CMV; cytomegalovirus; autologous; leukemia; hematological malignancies; stem cell transplantation; CMV reactivation; adoptive therapy
MeSH Terms: conditions — Leukemia; Hematologic Neoplasms | interventions — Leukapheresis; Blood Chemical Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Lymphopheresis — Lymphopheresis
Procedure: CMV specific lymphocyte infusion — CMV specific lymphocyte infusion
Procedure: Peripheral blood for CMV DNA PCR — Peripheral blood for CMV DNA PCR
Procedure: Haematology/Blood chemistry — Haematology/Blood chemistry analysis, Collection of blood for ancillary laboratory tests.

SUMMARY:
The investigators will assess whether the infusion of autologous CMV-specific T-cells at the time of CMV reactivation posttransplant will prevent worsening of CMV virus reactivation posttransplant to a level that warrants therapy with antiviral drugs (objectively assessed by looking at CMV virus copy number).

DETAILED DESCRIPTION:
Allogeneic Hematopoietic Stem Cell transplantation (allo-SCT) remains the only curative approach for a number of patients with hematological malignancies. However, the use of allo-SCT can expose patients to prolonged periods of immunosupression during which time viral infections can be a significant cause of morbidity and mortality.

Human cytomegalovirus (CMV) infection and reactivation still represents one of the most important and lifethreatening complications in immunocompromised patients. Prophylaxis or early treatment with antiviral drugs after CMV reactivation have reduced the mortality related to this complication. However, the antiviral drugs have many side-effects and are costly. Furthermore, CMV infection refractory to antiviral treatment after alloSCT is associated with a high mortality. A number of studies have shown the efficacy of selecting Tcells against the virus from the donor and infusing them into the recipient (adoptive transfer of immunity) to prevent or treat CMV reactivation. However this approach relies on the donor having preexisitng immunity to CMV (50% of the healthy population is CMV seronegative and therefore have no preexisting immunity against CMV). We propose an alternative approach to collect CMV specific Tcells from the seropositive recipient prior to transplantation; the autologous CMV specific T cells will then be infused back into the recipient at the time of CMV reactivation post-transplant.

This approach is especially relevant where the donor is CMV seronegative or unavailable or following the use of cord blood transplant where there is no memory T cell response to CMV.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received an allogeneic stem cell transplant from any donor, as treatment for a haematological malignancy.
2. HLAA0201 positive at one allele
3. CMV seropositive
4. The patient must be willing and capable of donating lymphocytes for CMVspecific CD8+ T cell selection using apheresis techniques
5. The patient must be in complete remission with no evidence of circulating blasts or other malignant cells
6. Patient must be fit to undergo leukapheresis
7. Patients must have signed an informed consent form before undergoing LP prior to alloSCT

Indications for infusion of autologous CMV specific CD8+ Tcells:

* Therapeutic: CMV disease following allogeneic stem cell transplantation
* Preemptive: CMV reactivation (by CMV DNA PCR)
* autologous CMV specific CD8+ T-cells must be infused into the patient no later than 72 following CMV reactivation.
* Steroids should be withdrawn at least 1 week before the infusion of CMVspecific CD8+ T-cell
* Patients must have signed an informed consent form before the infusion of autologous CMV specific CD8+ T-cells

Exclusion Criteria:

1. Patient CMV seronegative
2. No informed consent
3. Patient positive at the time of LP for one of the following infectious agents: HIV, HBV, HCV,Syphilis, HTLV 1 and 2
4. Patient with circulating leukemic blasts at the time of LP

Exclusion criteria for infusion of autologous CMV specific CD8+ T cells:

Severe GvHD (grade IIII-V) requiring full dose immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Response to adoptive transfer of autologous CMV-specific CD8+ T-cells | Up to three years
  Response to CMV-specific CD8+ T-cells administration will be measured and defined as a CMV DNA PCR< 50 copies.

SECONDARY OUTCOMES:
The occurrence of subsequent CMV reactivations | Up to three years
  The occurrence of subsequent CMV reactivations.
Rate of complete response | Up to three years
  The rate of complete response will be analyzed and compared to patients treated with anti-viral drugs only.
Rate of early complete response | Up to three years
  The rate of early complete response will be analyzed and compared to patients treated with anti-viral drugs only.
Rate of subsequent CMV reactivation | Up to three years
  The rate of subsequent CMV reactivation will be analyzed and compared to patients treated with anti-viral drugs only.

CONTACTS AND LOCATIONS:
Overall Officials: Katy Rezvani, MD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, London, United Kingdom